CLINICAL TRIAL: NCT05950529
Title: A Comparative, Randomized, Evaluator-Blind, Parallel-Group Clinical Study of the Effect of Two Experimental Lozenges on Oral Malodor After Single Use
Brief Title: Clinical Study of the Effect of Two Experimental Lozenges on Oral Malodor After Single Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novozymes A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NZ-OHBF-2020-01
Record Dates: First submitted 2023-07-11; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Oral Malodor
Keywords: enzymes, oral malodor
MeSH Terms: interventions — Flavoring Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Oral Malodor examiners are blinded and the subjects do not know which of the 2 lozenges they are taking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Experimental lozenge with the enzyme Polyphenol oxidase plus green coffee extract
  Interventions: Other: Experimental lozenge with the enzyme Polyphenol oxidase and green coffee extract
- Group B (Experimental): Experimental lozenge with the enzyme Polyphenol oxidase, green coffee extract and flavor
  Interventions: Other: Experimental lozenge with the enzyme Polyphenol oxidase, green coffee extract and flavor
- Group C (Placebo Comparator): Placebo lozenge Control (sorbitol only)
  Interventions: Other: Placebo lozenge control (sorbitol only)
- Group D (Other): No Product Control
  Interventions: Other: No product

INTERVENTIONS:
Other: Experimental lozenge with the enzyme Polyphenol oxidase and green coffee extract — Subjects will be instructed to allow their assigned lozenge to dissolve in the mouth while placed on the dorsal surface of the tongue. Subjects can suck on the lozenge and press the lozenge against the palate; however, the lozenge should not be moved around in the mouth or placed on the buccal mucosa. Subjects should avoid biting or chewing the lozenge and talking while dissolving the lozenge. After the lozenge has dissolved, the subject will be instructed to swallow the remaining solution.
  Arms: Group A
Other: Experimental lozenge with the enzyme Polyphenol oxidase, green coffee extract and flavor — Subjects will be instructed to allow their assigned lozenge to dissolve in the mouth while placed on the dorsal surface of the tongue. Subjects can suck on the lozenge and press the lozenge against the palate; however, the lozenge should not be moved around in the mouth or placed on the buccal mucosa. Subjects should avoid biting or chewing the lozenge and talking while dissolving the lozenge. After the lozenge has dissolved, the subject will be instructed to swallow the remaining solution.
  Arms: Group B
Other: Placebo lozenge control (sorbitol only) — Subjects will be instructed to allow their assigned lozenge to dissolve in the mouth while placed on the dorsal surface of the tongue. Subjects can suck on the lozenge and press the lozenge against the palate; however, the lozenge should not be moved around in the mouth or placed on the buccal mucosa. Subjects should avoid biting or chewing the lozenge and talking while dissolving the lozenge. After the lozenge has dissolved, the subject will be instructed to swallow the remaining solution.
  Arms: Group C
Other: No product — no product
  Arms: Group D

SUMMARY:
The goal of this clinical trial is to compare the control of oral malodor between an investigational lozenge with the enzyme polyphenol oxidase plus green coffee extract or an investigational lozenge with color and flavor along with the enzyme polyphenol oxidase plus green coffee extract in generally healthy subjects. Safety will be evaluated also.

Subjects will be randomly assigned to one of four study groups (group code: A, B, C or D):

* Experimental lozenge with the enzyme Polyphenol oxidase and green coffee extract
* Experimental lozenge with the enzyme Polyphenol oxidase, green coffee extract and flavor
* Placebo lozenge control (sorbitol only)
* No product control

Subjects will be asked to allow their assigned lozenge to dissolve in the mouth while placed on the dorsal surface of the tongue. Subjects can suck on the lozenge and press the lozenge against the palate; however, the lozenge should not be moved around in the mouth or placed on the buccal mucosa. Subjects should avoid biting or chewing the lozenge and talking while dissolving the lozenge. After the lozenge has completely dissolved, the subject will be instructed to swallow the remaining solution. Immediately (no later than 5 minutes) after subjects use their assigned lozenge product or no product, subjects will receive organoleptic assessments (OI) by the 4-5 trained judges and VSC readings (OralChroma readings). Organoleptic measurements (OI) will be repeated at 30 minutes, 1, 2, 3, and 4 hours following test product use or no test product use.

OralChroma measurements will be performed again after 30 minutes, 1, 2, 3, and 4 hours after test product use or no test product. Subjects will complete a post-product performance questionnaire after the 1-hour OI and OralChroma assessments have been administered. Following the 4-hour OralChroma assessment, each subject will receive a final oral soft and hard tissue exam for safety.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for study participation, subjects must meet the following criteria:

1. Generally healthy males and females ≥ 18 years of age.
2. Able to read, sign and receive a copy of the signed informed consent form.
3. Organoleptic score (Odor Intensity) ≥ 2 (morning breath: at least 6-12 hours following oral hygiene, eating or drinking) at Screening Visit, based on the average ratings of at least 4 Odor Intensity judges.
4. Have an OralChroma reading ≥ 125 ppb hydrogen sulfide H2S gas, vsc (at least 6-12 hours after eating or drinking or oral hygiene).
5. Intra-oral cause of bad breath (non-systemic origin) as determined by health history or exam.
6. Have at least 16 natural teeth.
7. Agree to abstain from eating, drinking, chewing gum, and any oral hygiene at least 6-12 hours prior to evaluation of oral malodor (Screening and Baseline visits).
8. Agree to avoid drinking alcohol beverages and eating spicy foods, garlic and onions, cabbage, spices, cauliflower and radishes (sulfur compounds) 48 hours prior to each study visit.
9. Agree to refrain from tongue brushing/cleaning for the duration of the study.
10. Adequate oral hygiene and no signs of oral neglect.
11. Has not taken any type of probiotic supplement intended for oral health within 14 days of screening visit.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. History of allergy or significant adverse effects following use of oral hygiene products such as toothpastes, mouth rinses, breath mints, lozenges, or chewing gum or their ingredients.
2. History of allergies to ingredients in the test product.
3. History of common food allergies (e.g. peanuts, tree nuts, milk, eggs, shellfish, fish, wheat, soybeans)
4. Self-reported as pregnant or nursing.
5. Self-reported serious medical conditions.
6. Based on history and clinical exam: advanced periodontitis, frank caries, and mucosal diseases.
7. Antibiotic or anti-inflammatory medication within 30 days of screening visit.
8. Dental prophylaxis or use of chemotherapeutic antiplaque/antigingivitis oral care products or tooth bleaching within 7 days of screening visit.
9. Smoker and/or user of smokeless tobacco products.
10. Orthodontic appliances, peri/oral piercings, or removable partial dentures.
11. Significant oral soft tissue pathology based on a visual examination.
12. Acute sinusitis or severe oral-pharyngeal infections.
13. Currently taking medications which can cause oral malodor.
14. Reduced salivary flow due to pathological reasons (e.g. Sjögrens syndrome).
15. Anything that, in the opinion of the investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study.
16. Participation in any oral care clinical study, concurrently or within the 30 days of screening exams.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Total VSC (OralChroma) readings | 5 minutes
  The mean total VSC (OralChroma) readings from the Baseline assessment to the immediate (5 minutes) assessment following product use.

SECONDARY OUTCOMES:
OI scores | 5 minutes, 30 minutes, 1, 2, 3, and 4 hours
  OI scores from the Baseline assessment (derived from mean odor ratings of the 4 judges) to immediate (5 minutes), 30 minutes, 1, 2, 3, and 4 hours following product use.
Total VSC (OralChroma) readings | 30 minutes, 1, 2, 3, and 4 hours
  Mean total VSC (OralChroma) readings from the Baseline assessment to assessments 30 minutes, 1, 2, 3, and 4 hours following product use.
Three major components of VSCs in mouth air | 5 minutes, 30 minutes, 1, 2, 3, and 4 hours
  Mean levels of each of the three major components of VSCs in mouth air: hydrogen sulfide (H2S), methyl mercaptan (CH3SH), and dimethyl sulfide ([CH3]2S) gases from the Baseline assessment to immediate (5 minutes), 1, 2, 3, and 4 hours following product use.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Milleman, DDS, MPA, Principal Investigator — Salus Research
Locations (1):
- Salus Research, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be kept confidential at the study center will not be shared externally.

REFERENCES:
- [Derived] Santos SL, Holz C, Milleman K, Milleman J, Wenqian G, Mateo LR. Effectiveness of a combination of laccase and green coffee extract on oral malodor: a comparative, randomized, controlled, evaluator-blind, parallel-group trial. J Breath Res. 2024 Nov 25;19(1). doi: 10.1088/1752-7163/ad8e7c. PMID 39496199